CLINICAL TRIAL: NCT02265718
Title: A Randomized, Double Blind, Placebo Controlled Trial To Study Difference In Cognitive Learning Associated With Repeated Self-administration Of Remote Computer Tablet-based Application Assessing Dual-task Performance Based On Amyloid Status In Healthy Elderly Volunteers
Brief Title: A Study To Evaluate The Difference In iPad-Based Cognitive Video Game (Akili Interactive's Project: EVO) Performance In Amyloid-Positive Versus Amyloid-Negative Healthy Elderly Volunteers
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A9001489
Record Dates: First submitted 2014-10-13; First posted 2014-10-16 (Estimated); Last update posted 2019-06-05 (Actual); Status verified 2019-06

CONDITIONS: Healthy
Keywords: Healthy; elderly volunteers
MeSH Terms: interventions — Methylphenidate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- (Amyloid Negative)
  Interventions: Drug: Ritalin; Drug: Placebo
- Amyloid Positive
  Interventions: Drug: Ritalin; Drug: Placebo

INTERVENTIONS:
Drug: Ritalin — 1 - 20 mg tablet taken once on Day 0 and taken once on Day 28
  Other Names: methylphenidate hydrochloride 20mg tablet taken once on day 0 and once on day 28
  Groups: (Amyloid Negative)
Drug: Placebo — 1 - matching tablet taken once on Day 0 and once on Day 28
  Other Names: matched placebo tablet taken once on day 0 and once on day 28
  Groups: (Amyloid Negative)
Drug: Ritalin — 1 - 20 mg tablet taken once on Day 0 and taken once on Day 28
  Other Names: methylphenidate hydrochloride 20mg tablet taken once on day 0 and once on day 28
  Groups: Amyloid Positive
Drug: Placebo — 1 - matching tablet taken once on Day 0 and once on Day 28
  Other Names: matched placebo tablet taken once on day 0 and once on day 28
  Groups: Amyloid Positive

SUMMARY:
The purpose of the study is to evaluate the difference in learning and performance measures associated with repeated use of an iPad video game (Akili Interactive's Project: EVO) in healthy elderly volunteers based on amyloid status.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females between the ages of 70 and 80.
* Subjects must have BMI of 17.5 to 32 kg/m2 and total body weight > 110 pounds.
* Acceptable screening MRI and PET scans that pass quality control requirements.

Exclusion Criteria:

* Co-morbid diagnosis of clinically documented Alzheimer's disease; - Significant cognitive impairment;
* MMSE (mini mental state examination) score <26

Ages: 70 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 97 (Actual)
Dates: Start 2014-09; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
divided attention performance | Day 0 - Day 28
  The difference in effect of cognitive training on divided attention performance as measured by teh pre/post training change in interference cost on EVO dueal task assessment at Day 28.

SECONDARY OUTCOMES:
sustained attention, impulsivity and episodic memory | Day 0 - Day 28
  The difference in effect of cognitive training on sustained attention, impulsivity and episodic memory as measured by the pre/post training change in performance at day 28
perforamce on EVO dual task assessment, TOVA and RAVLT | Day 0 - Day 28
  The performance on EVO dual task assessment, Test of Variables of Attention (TOVA and Rey Auditory Verbal Learning Test (RAVLT) as measured by the pre and post training scores at Day 0 and Day 28
within subject change on EVO, TOVA and RAVLT | Day 0 - Day 28
  The within subject change on EVO dual task assessment, TOVA and RAVLT between day -28 and Day 0.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (4):
- United States (4):
  - Collaborative Neuroscience Network, LLC, Long Beach, California
  - Broward Research Group, Hollywood, Florida
  - Miami Research Associates, South Miami, Florida
  - Jasper Clinic, Inc., Kalamazoo, Michigan

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A9001489&StudyName=A%20Study%20To%20Evaluate%20The%20Difference%20In%20iPad-Based%20Cognitive%20Video%20Game%20%28Akili%20Interactive%27s%20Project%3A%20EVO%29%20Performance%20In%20Amyloid-Posi